CLINICAL TRIAL: NCT06731894
Title: A Pilot Study to Evaluate the Benefits of Phytocannabinoids for the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Phytocannabinoids for Reducing Chronic Chemotherapy-Induced Peripheral Neuropathy in Breast and Colon Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24435; NCI-2024-08847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24435 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-12-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma; Chemotherapy-Induced Peripheral Neuropathy; Colon Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Specimen Handling; Cannabidiol; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Every bottle will be labelled in a blinded fashion. IDS Pharmacy will obtain the unblinded key. The study team, including the physician, will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (CBD) (Experimental): Patients receive CBD PO QD on days 1-3 of cycle 1, BID on days 4-6 of cycle 1, and TID on days 7-28 of cycle 1. Patients receive CBD PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.
  Interventions: Procedure: Biospecimen Collection; Drug: Cannabidiol; Other: Survey Administration
- Arm II (THC:CBD) (Experimental): Patients receive THC:CBD PO QD on days 1-3 of cycle 1, BID on days 4-6 of cycle 1, and TID on days 7-28 of cycle 1. Patients receive THC:CBD PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.
  Interventions: Procedure: Biospecimen Collection; Drug: Cannabidiol; Drug: Dronabinol; Drug: Placebo Administration; Other: Survey Administration
- Arm III (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-3 of cycle 1, BID on days 4-6 of cycle 1, and TID on days 7-28 of cycle 1. Patients receive placebo PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cannabidiol — Given PO
  Other Names: CBD; CBD Oil; Epidiolex; GWP42003-P
  Arms: Arm I (CBD); Arm II (THC:CBD)
Drug: Dronabinol — Given PO
  Other Names: (-)-.DELTA.9-Tetrahydrocannabinol; Abbott 40566; Delta(9)-Tetrahydrocannibinol; Delta-9-Tetrahydrocannabinol; Delta-9-THC; Delta9-THC; Marinol; SP 104; SP-104; SYNDROS; Tetrahydro-6,6,9-trimethyl-3-pentyl-6H-dibenzo(b,d)pyran-1-ol; Tetrahydrocannabinol; THC
  Arms: Arm II (THC:CBD)
Drug: Placebo Administration — Given PO
  Arms: Arm II (THC:CBD); Arm III (placebo)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trials evaluates how well different types of phytocannabinoids (cannabidiol [CBD] versus tetrahydrocannabinol [THC] and CBD formulation [THC:CBD]) work to reduce chronic chemotherapy-induced peripheral neuropathy among breast and colon cancer survivors. Chemotherapy induced peripheral neuropathy is a set of symptoms that includes pain, tingling, numbness and motor weakness caused by certain types of chemotherapy treatment. Phytocannabinoids are compounds made by the cannabis plant, such as THC and CBD, that have been found to be an effective treatment for chronic pain. Phytocannabinoids may be effective in reducing chronic chemotherapy-induced peripheral neuropathy symptoms in patients treated for breast or colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the ability of CBD and THC:CBD to reduce chronic chemotherapy-induced peripheral neuropathy (CIPN) symptoms as compared to placebo using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) among breast and colon cancer survivors.

SECONDARY OBJECTIVES:

I. Evaluate the impact of CBD and THC:CBD as compared to placebo on quality of life using the Functional Assessment of Cancer Therapy-General (FACT-G) among breast and colon cancer survivors with chronic CIPN.

II. Document the utilization of neuropathic and pain medications by cancer patients with chronic CIPN during treatment with CBD and THC:CBD as compared to placebo.

III. Describe the side effects of CBD and THC:CBD treatment.

EXPLORATORY OBJECTIVES:

I. Assess neurological symptoms and function with the Neuropathy Pain Scale (NPS), Total Neuropathy Score - Clinically Based (TNSc), Quantitative Sensory Testing (QST), Grooved Pegboard Test (GPT), Timed Up and Go (TUG) Test, and Unipedal Stance Balance Test (USBT) among patients with chronic CIPN treated with CBD and THC:CBD as compared to placebo.

II. Evaluate for predictors of response to CBD and THC:CBD for chronic CIPN.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive CBD orally (PO) once daily (QD) on days 1-3 of cycle 1, twice daily (BID) on days 4-6 of cycle 1, and three times daily (TID) on days 7-28 of cycle 1. Patients receive CBD PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.

ARM II: Patients receive THC:CBD PO QD on days 1-3 of cycle 1, BID on days 4-6 of cycle 1, and TID on days 7-28 of cycle 1. Patients receive THC:CBD PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.

ARM III: Patients receive placebo PO QD on days 1-3 of cycle 1, BID on days 4-6 of cycle 1, and TID on days 7-28 of cycle 1. Patients receive placebo PO TID on days 1-28 of cycle 2. Cycles repeat every 28 days for up to 2 cycles in the absence of unacceptable toxicity. Patients undergo urine collection during screening.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Willingness to comply with all study interventions including the use of medical cannabis and follow-up assessments
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group Performance Status Scale (ECOG) score ≤ 2
* Ability to read and understand English for questionnaires
* Patients must have either neuropathy ≥ 1 according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 scale or a neuropathy score of > 3 on a 0-10 scale plus a FACT/GOG-Ntx score of > 10
* The patient's previous chemotherapy treatment must have included a taxane (paclitaxel, nab-paclitaxel, or docetaxel) or platinum (cisplatin, oxaliplatin, or carboplatin) and considered the primary cause of the neuropathy by the medical team
* Total bilirubin ≤ 1.5 X upper limits of normal (ULN) (unless has Gilbert's disease) (To be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) ≤ 3 x ULN (To be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) ≤ 3 x ULN (To be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (To be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Current active treatment with chemotherapy, radiation or surgery in the past 3 months or planned treatment during this study protocol period. Note: Hormonal therapy is allowed
* Treatment with any neuropathic agent including taxane, platinum, vinca alkaloid, or bortezomib chemotherapy within the past 6 months
* Concurrent use of other alternative medicines such as medical cannabis, herbal agents and high dose vitamins and minerals
* Liver cirrhosis Child-Pugh B or C
* Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry. (These patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.)
* History of diabetic neuropathy, neuropathy related to HIV, or other medical causes of chronic neuropathy in the baseline assessment including past medical history, any history of diabetes, alcoholism, and vitamin B deficiency
* Previous medical cannabis use for any indication within 30 days of enrollment
* Planned or actual changes in type of medications that could affect symptoms related to CIPN. New medications for the treatment of CIPN are not allowed during the study.

  * Subjects need to be on stable doses of CIPN medications for 4 weeks
* Strong inhibitors or inducers of CYP3A4
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Diagnosis of Gilbert's disease
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* Patients who have an allergy or an aversion to strawberry or strawberry flavoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Subjectively experienced symptoms of peripheral neuropathy | Up to 28 days after last dose of therapy
  Assessed via Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity Subscale (FACT/GOG-Ntx). Will compare difference scores from the FACT/GOG-Ntx between all these groups using analysis of variance. A paired t-test will be utilized to compare scores between baseline and 8 and 12 weeks of treatment for each group separately.

SECONDARY OUTCOMES:
Health-related quality of life | Up to 28 days after last dose of therapy
  Assessed via Functional Assessment of Cancer Therapy-General. A paired T-test will be utilized to compare scores between baseline and 8 weeks of treatment. For comparisons between groups at four specific assessment points (baseline, week 4, week 8, and week 12), a repeated measures analysis of variance analysis will be performed.
Neuropathic medication utilization | Up to 28 days after last dose of therapy
  Neuropathic medication utilization data will initially be analyzed as a dichotomous variable (yes/no) for each medication. Comparisons between the baseline and after-treatment medication status will be analyzed using McNemar's test. Including all the time points in the analysis of any single medication will use Cochran's Q test.
Pain medication utilization | Up to 28 days after last dose of therapy
  Pain medication utilization data will initially be analyzed as a dichotomous variable (yes/no) for each medication. Comparisons between the baseline and after-treatment medication status will be analyzed using McNemar's test. Including all the time points in the analysis of any single medication will use Cochran's Q test.
Incidence of adverse events | Up to 28 days after last dose of therapy
  All adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 6.0. The severe adverse events (SAE) (grade ≥ 3) will be tabulated per treatment arm and the difference of SAE will be compared among groups using chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California